CLINICAL TRIAL: NCT00188448
Title: MRI of the Superficial Temporal Artery
Brief Title: MRI Superficial Temporal Artery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0223
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2005-09

CONDITIONS: Temporal Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

INTERVENTIONS:
Device: MRI

SUMMARY:
Repeat MRI of the Superficial temporal Artery in 5 volunteers

DETAILED DESCRIPTION:
Repeat MRI of the Superficial temporal Artery in 5 volunteers

ELIGIBILITY:
Inclusion Criteria:

* controls with normal temporal arteries

Exclusion Criteria:

* contraindication to MR

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 2003-04; Study Completion 2004-04

PRIMARY OUTCOMES:
Accuracy in displaying the superfifical temporal artery

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FRCP C, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada